CLINICAL TRIAL: NCT05047016
Title: A Virtual Clinical Trial to Implement and Evaluate the Dynamic Consent Model Based on the Blockchain-based Next-generation Clinical Trial Platform METORY
Brief Title: Study to Evaluate the Dynamic Consent Model Based on the Blockchain-based Clinical Trial Platform METORY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, SeungHwan Lee, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: METORY-101
Record Dates: First submitted 2021-09-08; First posted 2021-09-16 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-11

CONDITIONS: COVID-19 Pneumonia
Keywords: blockchain, dynamic consent

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dynamic consent arm (Other): Subjects will receive a virtual investigational product once daily. Subjects also need to measure their body temperature once daily at the scheduled timepoint.
  Interventions: Other: Virtual investigational product

INTERVENTIONS:
Other: Virtual investigational product — The virtual investigational product is a predefined text (e.g. AB123F). By entering the code into the application, the virtual 'administration' of the IP is conducted.

SUMMARY:
Blockchain technology has gained attention for its decentralized feature and data integrity. The study aims to apply blockchain technology to implement dynamic consent model and evaluate the real-world experience as a form of virtual clinical trial.

DETAILED DESCRIPTION:
The study will simulate a clinical trial that implements dynamic consent module. In this study, two major and three minor protocol amendments will be conducted on the scheduled date. Each subjects will give consent using the dynamic consent platform, METORY, and will be informed when the protocol is amended. The communication only be conducted under the METORY and the real-world experience of METORY would be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who can use METORY (application platform)
* Subjects who completely understand the study and voluntarily decide to participate in the study

Exclusion Criteria:

* Subjects who are not able to use the web or application due to cognitive dysfunction or other reasons
* Subjects who are not able to measure body temperature by themselves
* Subjects who investigators decide not be appropriate for the study for other reasons

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-09-13 (Actual); Primary Completion 2021-11 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Response time | Study Period of 4 weeks
  The time interval between notification of protocol amendment and subjects' response (consent)

SECONDARY OUTCOMES:
Study completion rate | Study Period of 4 weeks
  The proportion of subjects who completed the study
Dropout rate | Study Period of 4 weeks
  The proportion of subjects who withdrew the study

CONTACTS AND LOCATIONS:
Overall Officials: SeungHwan Lee, M.D., Ph.D., Principal Investigator — Seoul National University Hospital
Locations (2):
- South Korea (2):
  - Jeonbuk National University Hospital, Jeonju, Jeollabuk-do
  - Seoul National University Hospital, Seoul, Jongno-gu

IPD SHARING:
Plan to Share IPD: No